CLINICAL TRIAL: NCT05465096
Title: Interventional Pilot Study on the Treatment of Osteoarthritis of the Hip Joint With Intra-articular Ultrasound-guided Infiltration of Microfractured Autologous Adipose Tissue Containing Mesenchymal Stromal Cells
Brief Title: Treatment of Osteoarthritis of the Hip Joint With Intra-articular Injection of Microfractured Autologous Adipose Tissue Containing Mesenchymal Stromal Cells.
Acronym: Lipo-Hip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lipo-Hip
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Hip Osteoarthritis; Hip Disease
Keywords: MF-AT; MF-AT injection; Mesenchymal stromal cells; Pilot study; Hip; Micro-fragmented Adipose Tissue
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: Interventional pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MF-AT injection (Experimental): Patients will be treated with an intra-articular-ultrasound-guided injection of Micro-fragmented adipose tissue containing mesenchymal stromal cells.
  Interventions: Procedure: Micro-fragmented adipose tissue injection

INTERVENTIONS:
Procedure: Micro-fragmented adipose tissue injection — Intra-articular ultrasound-guided injection of MF-AT

SUMMARY:
The aim of the study is to evaluate the safety and efficacy up to 12 months of MF-AT in the echo-guided infiltrative treatment of hip OA through clinical, subjective and objective evaluations.

DETAILED DESCRIPTION:
For this pilot study, will be enrolled 30 patients with OA of the hip. All patients will be treated with a single infiltration of MF-AT obtained by the Lipogems® method. All activities of the present trial will be carried out at the Rizzoli Orthopaedic Institute (selection and enrollment, abdominal sampling, infiltrative treatment and follow-ups).

Patients will undergo infiltrative treatment after collecting informed consent for study participation and biographical data. Thereafter, patients will be followed up with clinical evaluation at 1-3-6-12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40 and 70 years;
2. Signs and symptoms of hip OA (pain intensity of at least 4 points and not more than 8 of VAS pain - 0-10 scale in the previous week);
3. Radiographic signs of hip OA (Grade 1-2 according to Tonnis classification) or MRI signs (chondropathy or minimal labrum degeneration without acute lesions) even if Grade 0.
4. Unilateral involvement;
5. Ability and consent of patients to actively participate in clinical follow-up;
6. Signature of informed consent.

Exclusion Criteria:

1. Patients unable to express consent;
2. Patients undergoing infiltration of other substance in the previous 6 months;
3. Patients undergoing lower limb surgery to be treated in the previous 12 months;
4. Patients with malignant neoplasms;
5. Patients with rheumatic diseases;
6. Patients with uncontrolled diabetes;
7. Patients with uncontrolled thyroid metabolic disorders;
8. Patients abusing alcoholic beverages, drugs or medications;
9. Body Mass Index > 35;
10. Pregnant and/or fertile women.
11. Pain intensity less than 4 points or greater than 8 in accordance with the VAS scale.
12. Patients with other hip pathologies: acetabular protrusion, concentric migration of the femoral head, presence of excessive deformity resulting from acetabular or femoral head dysplasia, collapse deformity, and deformed femoral head sequelae of Perthes disease or osteonecrosis of the femoral head.
13. Previous extensive surgery of the reference joint (osteotomy around the hip, open or arthroscopic osteochondroplasty for femoro-acetabular conflict).

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 6 months follow-up
  It's a standardized and widely used questionnaire to assess the condition of patients with osteoarthritis of the knee and includes assessment of pain, stiffness, and physical function of the joints. It can be administered to the patient.
  It measures 5 items for pain (range 0-20), two for stiffness (range 0-8), and 17 for functional limitation (range 0-68) that mainly relate to activities of daily living (e.g., getting up from a sitting position, bending over, going up and down stairs etc.); The score is then normalized on a 0-100 scale. Higher values indicate a worse outcome

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | baseline, 1 month, 3 months and 12 months follow-up
  It's a standardized and widely used questionnaire to assess the condition of patients with osteoarthritis of the knee and includes assessment of pain, stiffness, and physical function of the joints. It can be administered to the patient.
  It measures 5 items for pain (range 0-20), two for stiffness (range 0-8), and 17 for functional limitation (range 0-68) that mainly relate to activities of daily living (e.g., getting up from a sitting position, bending over, going up and down stairs etc.); The score is then normalized on a 0-100 scale. Higher values indicate a worse outcome
Visual Analogue Scale (VAS) | baseline, 1 month, 3 months, 6 months and 12 months follow-up
  VAS is a visual analogue scale consisting of a range scale (10 cm length), the ends of which correspond to "no pain" and "the strongest pain imaginable".
Harris Hip Scale (HHS) | baseline, 1 month, 3 months, 6 and 12 months follow-up
  This scale was developed for the evaluation of hip surgery outcomes and is intended to assess various hip disabilities and treatment methods in an adult population. The four sections that make up the questionnaire are: pain, function, absence of deformity, and range of motion. The HHS is a measure of dysfunction, so higher is the score, better is the outcome for the individual. The maximum possible score is 100.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Zaffagnini, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Filardo G, Perdisa F, Roffi A, Marcacci M, Kon E. Stem cells in articular cartilage regeneration. J Orthop Surg Res. 2016 Apr 12;11:42. doi: 10.1186/s13018-016-0378-x. PMID 27072345
- [Background] Tremolada C, Colombo V, Ventura C. Adipose Tissue and Mesenchymal Stem Cells: State of the Art and Lipogems(R) Technology Development. Curr Stem Cell Rep. 2016;2(3):304-312. doi: 10.1007/s40778-016-0053-5. Epub 2016 Jul 13. PMID 27547712
- [Background] Agarwal N, Mak C, Bojanic C, To K, Khan W. Meta-Analysis of Adipose Tissue Derived Cell-Based Therapy for the Treatment of Knee Osteoarthritis. Cells. 2021 Jun 1;10(6):1365. doi: 10.3390/cells10061365. PMID 34206010
- [Background] Meadows MC, Elisman K, Nho SJ, Mowry K, Safran MR. A Single Injection of Amniotic Suspension Allograft Is Safe and Effective for Treatment of Mild to Moderate Hip Osteoarthritis: A Prospective Study. Arthroscopy. 2022 Feb;38(2):325-331. doi: 10.1016/j.arthro.2021.04.034. Epub 2021 Apr 30. PMID 33940131
- [Background] Whitney KE, Briggs KK, Chamness C, Bolia IK, Huard J, Philippon MJ, Evans TA. Bone Marrow Concentrate Injection Treatment Improves Short-term Outcomes in Symptomatic Hip Osteoarthritis Patients: A Pilot Study. Orthop J Sports Med. 2020 Dec 9;8(12):2325967120966162. doi: 10.1177/2325967120966162. eCollection 2020 Dec. PMID 33344667
- [Background] Emadedin M, Ghorbani Liastani M, Fazeli R, Mohseni F, Moghadasali R, Mardpour S, Hosseini SE, Niknejadi M, Moeininia F, Aghahossein Fanni A, Baghban Eslaminejhad R, Vosough Dizaji A, Labibzadeh N, Mirazimi Bafghi A, Baharvand H, Aghdami N. Long-Term Follow-up of Intra-articular Injection of Autologous Mesenchymal Stem Cells in Patients with Knee, Ankle, or Hip Osteoarthritis. Arch Iran Med. 2015 Jun;18(6):336-44. PMID 26058927
- [Background] Mardones R, Jofre CM, Tobar L, Minguell JJ. Mesenchymal stem cell therapy in the treatment of hip osteoarthritis. J Hip Preserv Surg. 2017 Mar 19;4(2):159-163. doi: 10.1093/jhps/hnx011. eCollection 2017 Jul. PMID 28630737
- [Background] Rodriguez-Fontan F, Piuzzi NS, Kraeutler MJ, Pascual-Garrido C. Early Clinical Outcomes of Intra-Articular Injections of Bone Marrow Aspirate Concentrate for the Treatment of Early Osteoarthritis of the Hip and Knee: A Cohort Study. PM R. 2018 Dec;10(12):1353-1359. doi: 10.1016/j.pmrj.2018.05.016. Epub 2018 May 29. PMID 29857166
- [Background] Mikkelsen RK, Blond L, Holmich LR, Molgaard C, Troelsen A, Holmich P, Barfod KW. Treatment of osteoarthritis with autologous, micro-fragmented adipose tissue: a study protocol for a randomized controlled trial. Trials. 2021 Oct 27;22(1):748. doi: 10.1186/s13063-021-05628-4. PMID 34706757
- [Background] Pak J, Lee JH, Pak N, Pak Y, Park KS, Jeon JH, Jeong BC, Lee SH. Cartilage Regeneration in Humans with Adipose Tissue-Derived Stem Cells and Adipose Stromal Vascular Fraction Cells: Updated Status. Int J Mol Sci. 2018 Jul 23;19(7):2146. doi: 10.3390/ijms19072146. PMID 30041472